CLINICAL TRIAL: NCT02261233
Title: Osteopathic Manipulative Treatment and Postural Control: Systems Engineering Approach
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding for this project ended as of August 31, 2018
Sponsor: Michigan State University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jacek Cholewicki, Walter F. Patenge Professor, Michigan State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: NCCAM U19 AT006057 Project 1; 5U19AT006057-02 (NIH)
Record Dates: First submitted 2014-09-19; First posted 2014-10-10 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate treatment (Experimental): This arm receives osteopathic manipulative treatment shortly after enrollment
  Interventions: Procedure: Osteopathic manipulative treatment
- Delayed treatment (Experimental): This arm receives osteopathic manipulative treatment approximately 4 weeks after enrollment
  Interventions: Procedure: Osteopathic manipulative treatment

INTERVENTIONS:
Procedure: Osteopathic manipulative treatment — Up to 4 sessions of osteopathic manipulative treatment (once per week)

SUMMARY:
The overall goal of this project is to develop sensitive and objective clinical research tools for the assessment of postural control of the trunk. In order to accomplish this goal, we aim to quantify balance performance in an unstable seated task. Specifically, the investigators will quantify balance performance in low back pain participants before and after osteopathic manipulative treatment. The investigators hypothesize that there will be a significant improvement in balance performance after a single session of osteopathic manipulative treatment as well as after 4 sessions of osteopathic manipulative treatment and this improvement will be greater than any learning effect.

A secondary objective of this study is to quantify differences in patient-oriented outcome measures (e.g., self-reported pain, disability) in low back pain participants before and after osteopathic manipulative treatment. The investigators hypothesize that there will be a significant improvement in these self-reported outcomes following osteopathic manipulative treatment. The association between improvement in postural control parameters and patient-oriented measures will also be explored.

ELIGIBILITY:
Inclusion Criteria:

All participants must meet all of the inclusion criteria to participate in the study. Below is a list of inclusion criteria for LBP participants:

* Age 21-65 years
* Independently ambulatory
* Able to speak and read English
* Able to understand study procedures and to comply with them for the entire length of the study.
* Willing to be randomized to either immediate or delayed treatment group.
* Musculoskeletal pain - primarily in the low back region
* Pain rating equal to or greater than 3 out of10 as indicated on the Numeric Rating Scale for Pain
* Disability equal to or greater than 26% as indicated on the Oswestry Disability Questionnaire

Exclusion Criteria:

All candidates meeting any of the exclusion criteria at baseline will be excluded from study participation. Exclusion criteria will be self-reported. However, during each treatment session, the physicians will be watching for clinical signs and symptoms not consistent with physical findings that are suggestive of the presence of any of the exclusion criteria. In such a case, further treatment will be discontinued and the subject will be excluded.

Below is a list of exclusion criteria:

* Inability or unwillingness of individual to give written informed consent.
* Physical therapy or any other form of manual medicine (e.g., Osteopathic Manipulative Medicine, Chiropractic Manipulation, etc.), acupuncture or spinal injections within one month prior to study enrollment
* Workers' compensation benefits in the past 3 months or ongoing medical legal issues
* Possibly pregnant
* Obesity (BMI>32)
* Currently using electrical implants (e.g., cardiac pacemakers, drug delivery pumps, etc.)

History of:

* Spinal surgery
* Spinal fracture
* Spinal infection (e.g., osteomyelitis)
* Cancer

Unresolved symptoms from:

* Head trauma
* Inner ear infection with associated balance and coordination problems
* Orthostatic hypotension
* Uncontrolled hypertension
* Vestibular disorder (e.g. vertigo)

Current diagnosis of:

* Significant spinal deformity (e.g., scoliosis > 20 degrees, torticollis)
* Ankylosing spondylitis
* Spondylolisthesis grades III or IV
* Cauda equine syndrome
* Rheumatoid arthritis
* Osteoporosis
* Angina or congestive heart failure symptoms
* Active bleeding or infection in the back
* Blindness
* Seizures
* Neurologic disease (e.g., Parkinson's disease, multiple sclerosis, cerebral palsy, Alzheimer's disease, amyotrophic lateral sclerosis, stroke or transient ischemic attack in the past year, cervical dystonia)

Conditions recognized by a physician any time during the study:

* Significant or worsening signs of neurologic deficit
* Symptoms are not consistent with mechanical findings
* Other conditions impeding protocol implementation

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Change in postural control | Change from baseline to shortly after first treatment (1-2 days), from baseline to an expected average of week 4, and from week 4 to an expected average of week 8.
  Postural control will be assessed in an unstable seated task, in which subjects will be asked to balance on a specially designed seat. The average deviations from the neutral seat position will be measured in degrees.
Change in trunk muscle reflex latency | Change from baseline to shortly after first treatment (1-2 days), from baseline to an expected average of week 4, and from week 4 to an expected average of week 8.
  Subjects will be pulling with their trunk on a cable held by an electromagnet. The electromagnet will be suddenly released. Trunk muscle response to sudden load release will be measured on electromyographical recordings in milliseconds.

SECONDARY OUTCOMES:
Change in Patient Reported Outcomes Measurement Information System (PROMIS) | The expected average is weekly for this outcome measure until the end (expected average of 8 weeks).
  Assesses weekly changes in physical function, anxiety, depression, fatigue, sleep, satisfaction with social role, and pain with PROMIS-29 questionnaire.
Change in concomitant medication | The expected average is weekly for this outcome measure until the end (expected average of 8 weeks).tcome measure until the end, an expected average of 8 weeks.
  Assesses weekly changes in the use of medication for treating low back pain, including the type of medication and the quantity of medication (i.e., number of pills) with a questionnaire.
Change in Oswestry Disability Index | The expected average is weekly for this outcome measure until the end (expected average of 8 weeks).
  Assesses weekly changes in functional activities related to low back disability with the Oswestry Disability Index questionnaire.
Change in fear avoidance behavior | The expected average is weekly for this outcome measure until the end (expected average of 8 weeks).
  Assesses weekly changes in fear avoidance behavior using the Fear Avoidance Beliefs questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Cholewicki, PhD, Principal Investigator — Michigan State University; Norman P Reeves, PhD, Principal Investigator — Michigan State University
Locations (3):
- United States (3):
  - MSU Osteopathic Manipulative Medicine, East Lansing, Michigan
  - MSU Musculoskeletal Rehabilitation, Lansing, Michigan
  - Michigan State University Center for Orthopedic Research, Lansing, Michigan

REFERENCES:
- [Background] Radebold A, Cholewicki J, Polzhofer GK, Greene HS. Impaired postural control of the lumbar spine is associated with delayed muscle response times in patients with chronic idiopathic low back pain. Spine (Phila Pa 1976). 2001 Apr 1;26(7):724-30. doi: 10.1097/00007632-200104010-00004. PMID 11295888
- See also: Website for Michigan State University Center for Orthopedic Research — http://orthopedicresearch.msu.edu/
- See also: Website for the National Center for Complementary and Alternative Medicine (Sponsor) — http://nccam.nih.gov/